CLINICAL TRIAL: NCT05357287
Title: Closed Incisional Negative Pressure Wound Therapy in Post-surgical Wound Care of Patients With Periprosthetic Joint Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMRPG3L1721
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-03

CONDITIONS: Wound Heal; Periprosthetic Joint Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevena (Experimental)
  Interventions: Device: PREVENA incision management system

INTERVENTIONS:
Device: PREVENA incision management system — We will apply Prevena on the surgical wound right after closure of the wound in the operating theater. Prevena will be used for 7 days, unless there is ongoing infection or much wound drainage that requires debridement.

SUMMARY:
In the proposed study, we will apply Prevena on the surgical wound right after closure of the wound in the operating theater. Prevena will be used for 7 days, unless there is ongoing infection or much wound drainage that requires debridement.

Most periprosthetic joint infections are from hematogenous origin. Hence, it is considered clean wound unless there is a discharging sinus.

ELIGIBILITY:
Inclusion Criteria:

1. patients with periprosthetic joint infection
2. indicated for debridement surgery
3. high risk for wound complication, including one of the followings: diabetes mellitus, use anticoagulants other than aspirin, current smoker, on immunomodulators or steroids, malnutrition, liver disease, renal failure, BMI > 35 kg/m2

Exclusion Criteria:

1. previous flap surgery on the indexed joint
2. younger than 18 years of age
3. silver allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
wound complication | 12 weeks
  Wound complication, including: Persistent wound drainage, blisters, hematoma, wound dehiscence, skin necrosis, suture abscess, cellulitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan